CLINICAL TRIAL: NCT07147465
Title: Indicateurs de Performance et Impact Sur le Parcours de Soins du Séquençage Sur Les Plateformes Seqoia et Auragen (Seqogen) Pour Les Patients en Oncologie
Brief Title: Performance Indicators and Impact on the Care Pathway of Sequencing on the SeqOIA and AURAGEN (Seqogen) Platforms for Oncology Patients
Acronym: SONCO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: AuraGen Aesthetics LLC (Industry); Centre Leon Berard (Other); Laboratoire SeqOIA (Unknown); PLAN FRANCE MÉDECINE GÉNOMIQUE 2025 (Unknown)
Responsible Party: Sponsor
Other Study IDs: AP-HP
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-07

CONDITIONS: Cancer; NGS; Tumor; RARE DISEASE
Keywords: Oncology; genomic medecine; cancer; rare diseases; next-generation sequencing
MeSH Terms: conditions — Neoplasms; Rare Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
As part of the French Genomic Medicine Plan 2025 (FGM), the SeqOIA and AURAGEN platforms were selected to perform high-throughput genomic sequencing.

The SONCO (Sequencing Oncology Cohort) project combines their medical and economic evaluations into a single national cohort. Its objective is to assess the impact of genomic sequencing on care pathways and treatment recommendations by collecting indicators related to quality, turnaround time, and patient information. Clinical data are gathered from molecular tumor board reports (via SPICE and HYGEN) and from hospital medical records.

This cohort is intended to support public health decision-making and help anticipate the organization of future genomic platforms.

DETAILED DESCRIPTION:
SONCO is an observational cohort study designed to assess the clinical and organizational impact of implementing genomic sequencing in oncology. It collects data from all patients referred to either of the two platforms AURAGEN and SeqOIA, focusing on several key indicators: turnaround times, quality of patient information, and overall quality of care.

The study incorporates: Clinical and molecular decisions from national molecular tumor boards (MTB), recorded via digital tools such as SPICE and HYGEN; Additional clinical data from patient medical records before and after sequencing, collected from the hospitals where patients are followed.

The overarching aim is to evaluate how genomic information influences patient care trajectories and treatment decisions. By analyzing these real-world data, SONCO will contribute to optimizing future genomic medicine workflows, contribute to the development of national guidelines in partnership with professional societies, and help shape public health strategies. It also plays a critical role in anticipating the organizational and resource needs for scaling up genomic services across France.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer and referred for high-throughput sequencing
* Sequencing pre-indication validated: Patients for whom the pre-indication for sequencing the genome, exome, and RNA has been validated by the upstream RCP (Multidisciplinary Tumor Board) since January 1, 2021.

Consent for data reuse: Patients who have agreed to the reuse of their medical and genomic data for research purposes and have not opposed this use.

Exclusion Criteria:

* Opposition to data reuse, unvalidated upstream RCP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with cancer and referred for high-throughput sequencing
Sampling Method: Non-Probability Sample
Enrollment: 3149 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Calculation of result turnaround time. | 8 Weeks
  interval from the upstream Multidisciplinary Team (MDT) meeting to the downstream multidisciplinary meeting
Treatment recommendation issued following the downstream multidisciplinary meeting | 6 months
  Prescription details include the actual treatment prescribed, the patient's response to treatment, the number of therapy lines received after the initial prescription, the specific molecule prescribed, and the type of genomic alteration guiding the therapeutic choice.

SECONDARY OUTCOMES:
Sample Arrival Time for Analysis | 8 weeks
  Interval between the date of the upstream Multidisciplinary Team (MDT) meeting and the date of arrival of the tumor sample at one of the platforms for anatomical pathology prequalification/qualification
Elapsed time from sequencing to the signing of the medical biology report by the biologist | 8 Weeks
  Delay between the date of sequencing and the date the medical biology report is validated by the biologist.
Elapsed time from sequencing to the downstream multidisciplinary meeting. | 8 weeks
  Delay between the sequencing date and the downstream multidisciplinary meeting

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle DURAND-ZALESKI, Professor, Principal Investigator — Greater Paris University Hospitals
Locations (3):
- France (3):
  - Centre Leon Berard, Lyon
  - APHP Hôtel Dieu URC Economie de la sante /URC ECO, Paris
  - HOPITAL AP-HP Cochin, Paris